CLINICAL TRIAL: NCT00798057
Title: Clinical Outcomes Study of Proton Radiation Therapy for Pituitary Adenoma
Brief Title: Proton Radiation Therapy for Pituitary Adenoma
Acronym: PI01
Status: Terminated | Type: Observational
Why Stopped: Due to slow enrollment and feasibility issues.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 0701-PI01
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Pituitary Adenoma
Keywords: Pituitary tumor; Outcomes; Proton radiation
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Proton Radiation

SUMMARY:
The purpose of this study is to collect information from medical records to see what effects proton beam radiation has on pituitary tumors and analyze possible side effects.

DETAILED DESCRIPTION:
Data collection will be obtained from the patient's medical records including initial evaluation, pathology report, dosimetry information, radiotherapy completion records and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven pituitary adenoma.
* Age 18 years or older.
* Status post biopsy, gross total resection (from initial surgery for recurrent disease) or subtotal resection.
* Good to moderate neurological function status

Exclusion Criteria:

*Previous radiation that would compromise the ability to deliver the prescribed treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at a radiation oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Collect and analyze outcome data on tumor control. | When each patient has been followed for a minimum or 12 months and then again after 24 months to a maximum of 10 years.

SECONDARY OUTCOMES:
Collect and analyze outcome data on normal tissue morbidity. | When each patient has been followed for a minimum of 12 months and then again after 24 months to a maximum of 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ronny L Rotondo, MD, CM, FRCPC, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] Ezzat S, Asa SL, Couldwell WT, Barr CE, Dodge WE, Vance ML, McCutcheon IE. The prevalence of pituitary adenomas: a systematic review. Cancer. 2004 Aug 1;101(3):613-9. doi: 10.1002/cncr.20412. PMID 15274075
- [Background] Surawicz TS, McCarthy BJ, Kupelian V, Jukich PJ, Bruner JM, Davis FG. Descriptive epidemiology of primary brain and CNS tumors: results from the Central Brain Tumor Registry of the United States, 1990-1994. Neuro Oncol. 1999 Jan;1(1):14-25. doi: 10.1093/neuonc/1.1.14. PMID 11554386
- [Background] Turner HE, Stratton IM, Byrne JV, Adams CB, Wass JA. Audit of selected patients with nonfunctioning pituitary adenomas treated without irradiation - a follow-up study. Clin Endocrinol (Oxf). 1999 Sep;51(3):281-4. doi: 10.1046/j.1365-2265.1999.00865.x. PMID 10469006
- [Background] Brada M, Rajan B, Traish D, Ashley S, Holmes-Sellors PJ, Nussey S, Uttley D. The long-term efficacy of conservative surgery and radiotherapy in the control of pituitary adenomas. Clin Endocrinol (Oxf). 1993 Jun;38(6):571-8. doi: 10.1111/j.1365-2265.1993.tb02137.x. PMID 8334743
- [Background] Milker-Zabel S, Debus J, Thilmann C, Schlegel W, Wannenmacher M. Fractionated stereotactically guided radiotherapy and radiosurgery in the treatment of functional and nonfunctional adenomas of the pituitary gland. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1279-86. doi: 10.1016/s0360-3016(01)01535-8. PMID 11483339
- [Background] Stieber V, Deguzman A, et al. Pituitary. In: Perez CA, Brady LW, Halperin EC, Schmidt-Ullrich RK, editors. Principles and practice of radiation oncology. Philadelphia: Lippincott Williams and Wilkins; 2004. p.839-859.
- [Background] Minniti G, Traish D, Ashley S, Gonsalves A, Brada M. Risk of second brain tumor after conservative surgery and radiotherapy for pituitary adenoma: update after an additional 10 years. J Clin Endocrinol Metab. 2005 Feb;90(2):800-4. doi: 10.1210/jc.2004-1152. Epub 2004 Nov 23. PMID 15562021
- [Background] Bolsi A, Fogliata A, Cozzi L. Radiotherapy of small intracranial tumours with different advanced techniques using photon and proton beams: a treatment planning study. Radiother Oncol. 2003 Jul;68(1):1-14. doi: 10.1016/s0167-8140(03)00117-8. PMID 12885446
- [Background] Cozzi L, Fogliata A, Lomax A, Bolsi A. A treatment planning comparison of 3D conformal therapy, intensity modulated photon therapy and proton therapy for treatment of advanced head and neck tumours. Radiother Oncol. 2001 Dec;61(3):287-97. doi: 10.1016/s0167-8140(01)00403-0. PMID 11730999
- [Background] Cozzi L, Clivio A, Vanetti E, Nicolini G, Fogliata A. Comparative planning study for proton radiotherapy of benign brain tumors. Strahlenther Onkol. 2006 Jul;182(7):376-81. doi: 10.1007/s00066-006-1500-5. PMID 16826355